CLINICAL TRIAL: NCT07102758
Title: Evaluation of Soft and Hard Tissue Augmentation by Connective Tissue Graft or Leukocyte-Platelet Rich Fibrin in Immediate Implant Placement With Customized Healing Abutment: A Randomized Controlled Clinical Trial.
Brief Title: L-PRF vs Connective Tissue With Customized Healing Abutment in Immediate Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Salem, General dentist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-436
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Recession, Gingival; Bone Loss in Jaw
Keywords: L-prf; connective tissue; customized healing abutment; implant
MeSH Terms: conditions — Gingival Recession | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue with dental implant and customized healing abutment (Active Comparator): Connective tissue with dental implant and customized healing abutment
  Interventions: Procedure: Connective tissue with dental implant and customized healing abutment
- L-PRF with dental implant and customized healing abutment (Experimental): L-PRF with dental implant and customized healing abutment
  Interventions: Procedure: L-PRF with dental implant and customized healing abutment

INTERVENTIONS:
Procedure: L-PRF with dental implant and customized healing abutment — L-PRF with dental implant and customized healing abutment
  Arms: L-PRF with dental implant and customized healing abutment
Procedure: Connective tissue with dental implant and customized healing abutment — Connective tissue with dental implant and customized healing abutment
  Arms: Connective tissue with dental implant and customized healing abutment

SUMMARY:
comparison between L-prf and connective tissue with dental implant

DETAILED DESCRIPTION:
comparison between L-PRF and Connective tissue with customized healing abutment regaring soft and hard tissue outcomes with immediate dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Intact labial/buccal bone plate
* The presence of non-restorable single-rooted maxillary centrals, canines or premolars.
* Sufficient bone volume.
* Good oral hygiene.
* Nonsmokers.
* Sufficient bone width (≥ 1 mm) in the buccal plate of the remaining bone to place an implant confirmed by cone beam computer tomography (CBCT).

Exclusion Criteria:

* Insufficient bone volume.
* Active infection.
* Patients on chemotherapy or radiotherapy.
* Patients who have systemic disorders {uncontrolled diabetes mellitus, autoimmune disease, …etc},
* Pregnant patients,
* Patients with bone diseases
* Presence of periapical pathology.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Patient-reported pain experience | first 7 days after surgery
  Pain experience after surgery is daily measured by the patients using a visual analogue scale (VAS) in the first postoperative 7 days, with Day 0 being the day of the surgery. Before going to sleep, patients will be asked to mark the VAS that best represented the average pain they had experienced during the day.
Pink aesthetic score | before surgery, 3 months and 6 months after surgery
  Parameters are : 0,1 and 2.
  Mesial papilla : 0 ( Missing ) , 1 ( Incomplete ) and 2 ( Complete ).
  Distal Papilla : 0 ( Missing ) , 1 ( Incomplete ) and 2 ( Complete ).
  Tissue contour : 0 ( Unnatural) , 1 ( virtually natural ) and 2 ( natural).
  Gingival level : 0 ( >2mm) , 1 ( 1-2mm ) and 2 ( 1 mm).
  Alveolar process : 0 ( clearly resorbed ) , 1 ( slightly resorbed ) and 2 ( no difference).
  Coloring : 0 ( clear difference ) , 1 ( slight difference ) and 2 ( no difference).
  Texture : 0 ( clear difference ) , 1 ( slight difference ) and 2 ( no difference).
crestal bone loss | preoperative and 6 months post operative
  distance from implant shoulder to marginal bone

SECONDARY OUTCOMES:
Gingival thickness | pre opearative, 3 and 6 months post operative
  1 mm apical to gingival margin in mid buccal
probing pocket depth | preoperative , 3 and 6 months post operative
  mid buccal , mesio buccal , disto buccal and mid palatal
keratinized tissue width | preoperative , 3 and 6 months post operative
  in mid buccal, from gingival margin to mucogingival junction

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt